CLINICAL TRIAL: NCT01811355
Title: Mexiletine for the Treatment of Muscle Cramps in ALS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bjorn Oskarsson, MD (Other)
Collaborators: University of California, Davis (Other); ALS Association (Other)
Responsible Party: Sponsor-Investigator, Bjorn Oskarsson, MD, Assistant Professor of Clinical Neurology, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 378164
Record Dates: First submitted 2013-03-06; First posted 2013-03-14 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Muscle Cramps in Amyotrophic Lateral Sclerosis
Keywords: Muscle cramps; Cramp; ALS; Amyotrophic Lateral Sclerosis; Lou Gehrig's disease; Motor Neuron Disease; MND
MeSH Terms: conditions — Muscle Cramp; Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Mexiletine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mexiletine (Active Comparator): Mexiletine, capsule, 150mg, PO BID, 14 days
  Interventions: Drug: Mexiletine
- Placebo (Placebo Comparator): Placebo, capsule, PO BID, 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mexiletine — Sodium channel blocker
  Other Names: Mexetil
  Arms: Mexiletine
Drug: Placebo — Placebo
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if mexiletine is effective for the treatment of muscle cramps in Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
Background:

Many ALS patients suffer from painful muscle cramps, but unfortunately we do not have any medication proven to help muscle cramps in ALS. Reducing the pain caused by cramps - which can be debilitating - could help people living with ALS.

Muscle cramps are sudden, painful, and involuntary contractions of a muscle. They are caused by nerve dysfunction. When we examine nerves and muscles electrically, we see cramps as bursts of high-frequency (up to150 Hz) firing of the motor nerve cells. Cramps in ALS are believed to be the result of an increase of persistent sodium currents in the sick lower motor nerve cells.

A medication called Quinine was for many years the commonly used drug for controlling cramps in ALS, but the FDA has advised against its use for cramps because of its potential risks (e.g., death). Today there is no agreement on how to treat cramps in the ALS. The American Academy of Neurology recently encouraged further studies of the treatment of muscle cramps and suggested lidocaine as one of a few drugs of special interest.

Mexiletine:

Mexiletine is a medication closely related to lidocaine that can be taken by mouth (instead of being injected). Mexiletine stops the type of sodium currents that are thought to cause muscle cramps. Mexiletine is a relatively older medication that has been extensively studied in humans. It has been shown to reduce the electrical measures of muscle cramps for other disease conditions. For example, in patients with another severe nerve disease - Machado-Joseph disease (SCA3) - mexiletine treatment led to a decrease in the average number of muscle cramps from 24 to 3 cramps per month.. The safety profile of mexiletine is good, with the most frequent side effects being nausea or other abdominal symptoms. These side effects are rare at the doses (300 mg/day) used in this study. In patients with normal heart function, mexiletine has a minimal effect on heart rhythm. In previous clinical trials, no subject developed any serious heart rate problem.

Experimental Plan:

Using multiple sites within the State of California we will quickly enroll a small number (N=30) of ALS patients with severe muscle cramps. The study is a double-blinded, placebo controlled (i.e., the investigator and the participant does not know if the pills contain mexiletine or placebo), crossover (all subjects receive two weeks of mexiletine and two weeks of placebo) study.

After a one week run in, participants will be evaluated on their ability to fill out the cramp diary. Participants who filled out their diary will be randomly assigned to either mexiletine or placebo for their first two weeks. For the first three days of each 2-week period, one 150mg capsule will be taken at bed time. For day 4 to 14 one capsule twice per day will be taken. Each treatment period will be 2 weeks with an intervening 1 week washout period - for a total study length of 6 weeks. Safety will be monitored with liver function studies and EKG's.

ELIGIBILITY:
Inclusion Criteria:

* ALS diagnosed according to El Escorial criteria (Awaji version) as: Possible, Probable, or Definite.
* Experiencing cramps as a moderate or severe symptom as defined by willingness to take a medication for the symptom
* ≥2 cramps per week during run in week
* Life expectancy > 6 months, estimated by clinician
* Able to take drug capsule by mouth
* No significant EKG abnormality on screening
* aspartate aminotransferase / alanine aminotransferase <2x upper limit of normal measured at screening
* Having successfully filled out the cramp diary and cramp and fasciculation scales on six out of the last seven days of run in period

Exclusion Criteria:

* Inability to communicate by telephone or email
* Allergy/ known sensitivity to mexiletine
* Prior use of mexiletine
* AV block unless subject has pacemaker
* Cardiac arrhythmia
* Prior myocardial infarction
* Other significant EKG abnormality
* Liver disease
* History of leucopenia (WBC <3,500/mm3)
* Epilepsy
* Other serious and unstable medical condition
* Pregnant woman
* Breastfeeding woman
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Use of quinidine (alone or as a component of Nuedexta®) during the study
* Inability or unwillingness of subject to give written informed consent
* Woman of childbearing potential, not willing to use at least two approved methods of contraception
* Use of a prohibited medication during study

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Oskarsson, MD, Principal Investigator — UC Davis
Locations (6):
- United States (6):
  - UCD Telehealth Network - Lake Almanor Clinic, Chester, California
  - UCSD Department of Neurosciences ALS Clinical Trials (ACT) Program, La Jolla, California
  - UCLA Neuromuscular Research Program, Los Angeles, California
  - UCD Telehealth Network, Multiple Locations, California
  - UC Irvine Health ALS & Neuromuscular Center, Orange, California
  - UC, Davis Medical Center ALS Clinic, Sacramento, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 28 patients who signed consent, 5 did not meet inclusion criteria because of past myocardial infarction (n=1), long QT syndrome (n=1), AV block (n=1), no muscle cramps (n=1), and hospitalization during the screening period that resulted in inability to complete a screening diary and follow-up (n=1) .
Groups:
- Mexiletine First/Placebo Second: Mexiletine, capsule, 150mg, PO BID, 14 days
  Placebo, capsule, PO BID, 14 days
- Placebo First/Mexiletine Second: Placebo, capsule, PO BID, 14 days
  Mexiletine, capsule, 150mg, PO BID, 14 days
Period: First Dose
Arm/Group | Mexiletine First/Placebo Second | Placebo First/Mexiletine Second
Started | 11 | 12
Completed | 9 | 12
Not Completed | 2 | 0
Period: Washout
Arm/Group | Mexiletine First/Placebo Second | Placebo First/Mexiletine Second
Started | 9 | 12
Completed | 9 | 12
Not Completed | 0 | 0
Period: Second Dose
Arm/Group | Mexiletine First/Placebo Second | Placebo First/Mexiletine Second
Started | 9 | 12
Completed | 9 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Subjects Enrolled: A total of 23 subjects were enrolled. 11 were randomized to receive study drug first, followed by placebo. 12 subjects received placebo first and study drug second. Overall participant characteristics are displayed in the baseline table.
Arm/Group | Total Subjects Enrolled
Number analyzed (Participants) | 23
Age, Customized [Mean (Standard Deviation); unit: years]
  Years | 62.4 (12.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  males | 15
  females | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Daily Muscle Cramps
Description: The average of the daily recording of number of muscle cramps that occurred in the last 24 hours- over a 6 week period.
Time Frame: 6 weeks
Population: Among the 21 patients who completed the study, 1 patient did not return the outcome diary, which resulted in 20 patients available for analysis.
Measure: Mean (Standard Deviation); unit: Cramps per 24 hours
Arm/Group | Mexiletine First/Placebo Second | Placebo First/Mexiletine Second
Number analyzed (Participants) | 8 | 12
Cramps per 24 hours
  Placebo Dose | 6.1 (8.1) | 4.7 (4.2)
  Mexiletine Dose | 4.9 (8.0) | 2.5 (2.8)
  Difference Between | 1.2 (2.9) | 2.2 (2.2)

2. Primary Outcome: Cramp Severity
Description: Daily cramp severity was rated on the 100-unit visual analog scale. Scores ranged from 0 to 100, with 100 being the greatest amount of cramp severity
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mexiletine First: Mexiletine, capsule, 150mg, PO BID, 14 days
  Mexiletine: Sodium channel blocker
- Placebo First: Placebo, capsule, PO BID, 14 days
  Placebo: Placebo
Arm/Group | Mexiletine First | Placebo First
Number analyzed (Participants) | 8 | 12
units on a scale
  Placebo Dose | 43.6 (31.0) | 44.7 (26.7)
  Mexiletine Dose | 23.1 (16.8) | 32.8 (27.7)
  Difference Between | 20.5 (40.6) | 12.0 (18.1)

ADVERSE EVENTS:
Arm/Group | Mexiletine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 9/23 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mexiletine (N=23) | Placebo (N=21)
Dizzines (Nervous system disorders) | 1 (1) | 0 (0) — Mild
Fall (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) — Mild
Congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Mild
Chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Mild
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) — Mild
Increased urination (Renal and urinary disorders) | 1 (1) | 0 (0) — Mild
Itchiness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Mild
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No